CLINICAL TRIAL: NCT05271123
Title: Pulmonary Functions in Relation to Gross Motor Function Level in The Children With Cerebral Palsy
Brief Title: Pulmonary Functions in Relation to Gross Motor Function Level
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Abbass, Dr.Mai Elsayed Abbass, Lecturer of pediatric physical therapy, Cairo University
Other Study IDs: REC/012/003541
Record Dates: First submitted 2022-02-13; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Children were evaluated using spirometer to assess forced expiratory volume at first second and peak expiratory flow and gross motor function classification system to assess the functional level.
  Interventions: Diagnostic Test: Assessment of respiratory function and growth motor function classiffication level

INTERVENTIONS:
Diagnostic Test: Assessment of respiratory function and growth motor function classiffication level — Assessment of respiratory function using spirometer and assessment of growth motor function classiffication level using GMFCs

SUMMARY:
Aim: To investigate the relation between forced expiratory volume at first second and peak expiratory flow with gross motor function level in the children with cerebral palsy.

Methods and Procedures: Thirty children with cerebral palsy from both sexes were included in this study. The children ages ranged from 3 to 11 years old.

DETAILED DESCRIPTION:
Methods and Procedures: Thirty children with cerebral palsy from both sexes were included in this study. The children ages ranged from 3 to 11 years old. Children were evaluated using spirometer to assess forced expiratory volume at first second and peak expiratory flow and gross motor function classification system to assess the functional level.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* age was from 3 to 11years old
* They were able to sit independently and to follow instructions.
* Children who can blow air independently.

Exclusion Criteria:

* Uncontrolled convulsions
* Any psychiatric disorders

Ages: 3 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: * Children with cerebral palsy
  * age was from 3 to 11years old
  * They were able to sit independently and to follow instructions
  * Children who can blow air independently.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
FEV1 | baseline ( enrolment)
  Forced expiratory volume at first second
PEF | baseline ( enrolment)
  Peak Expiratory Flow Peak expiratory flow
GMFCs | baseline ( enrolment)
  Growth motor functional classification level

CONTACTS AND LOCATIONS:
Overall Officials: Mai Abbass, Ph.D., Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt